CLINICAL TRIAL: NCT07103980
Title: Inhaled Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Post-Infectious Cough: A Single-Center Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR-31-25-044025
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Post-Infectious Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell-derived exosomes and conventional treatment group (Experimental): Mesenchymal stem cell derived exosome nebulization (FITCELL 5ml nebulization QD) was combined with compound methoxyphenamine capsule ( "Asmei" 2 capsules oral TID) for cough treatment.
  Interventions: Drug: Mesenchymal stem cell derived exosome nebulization combined with compound methoxyphenamine capsule
- Placebo and conventional treatment group (Placebo Comparator): Normal saline nebulization (0.9% sodium chloride 5ml nebulization QD) was combined with the compound methoxyphenamine capsule ("Asmei" 2 capsules oral TID) for cough treatment.
  Interventions: Drug: Normal saline nebulization combined with the compound methoxyphenamine capsule

INTERVENTIONS:
Drug: Mesenchymal stem cell derived exosome nebulization combined with compound methoxyphenamine capsule — Mesenchymal stem cell derived exosome nebulization (FITCELL 5ml nebulization QD) was combined with compound methoxyphenamine capsule ( "Asmei" 2 capsules oral TID) for cough treatment.
  Arms: Mesenchymal stem cell-derived exosomes and conventional treatment group
Drug: Normal saline nebulization combined with the compound methoxyphenamine capsule — Normal saline nebulization (0.9% sodium chloride 5ml nebulization QD) was combined with the compound methoxyphenamine capsule ("Asmei" 2 capsules oral TID) for cough treatment.
  Arms: Placebo and conventional treatment group

SUMMARY:
This study is an exploratory clinical trial. It is intended to investigate the efficacy of mesenchymal stem cell-derived exosome nebulization in the treatment of postinfectious cough through a randomized controlled clinical study, with a view to providing better treatment options for patients with postinfectious cough, improving their quality of life, and providing reference data for the subsequent multi-center clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-60 years.
2. Diagnosis of post-infectious cough, which is defined as: after the symptoms of acute respiratory infection have disappeared, chest radiographs are normal, irritating dry cough or cough with small amounts of mucoid phlegm occurs, cough persists for 3 to 8 weeks, and other causes of cough are ruled out.
3. Baseline cough visual analog scale>=60mm.

Exclusion Criteria:

1. patients with any other disease that causes coughing (eg, Upper airway cough syndrome, eosinophilic bronchitis, gastroesophageal reflux cough, bronchial asthma, chronic obstructive pulmonary disease and bronchiectasis).
2. Patients with serious lung diseases (eg, lung cancer, tuberculosis or pulmonary fibrosis).
3. Patients with serious comorbidities, (eg, cardiovascular, cerebrovascular, liver, kidney or hematopoietic system diseases or other serious primary diseases)
4. Current or ex-smokers quitting smoking for less than 6 months.
5. Patients with a body temperature ≥37.3℃.
6. Patients with white blood cell count or neutrophil count is higher than the upper limit of normal.
7. Patients with abnormal chest X-rays.
8. Patients Suspected or confirmed history of alcohol or drug abuse or mental illness.
9. Patients with pregnancy, lactation or planning pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The change value of Leicester cough questionnaire | Day 7 of treatment initiation
  The primary endpoint of the study is the statistical difference in the absolute value of changes in the Leicester Cough Questionnaire (LCQ) score from baseline to Day 7 of treatment between the two groups of patients.

SECONDARY OUTCOMES:
The change value of Leicester cough questionnaire | Day 14 of treatment initiation
  The secondary endpoint of the study is the statistical difference in the absolute value of changes in the Leicester Cough Questionnaire (LCQ) score from baseline to Day 14 of treatment between the two groups of patients.
The change value of cough symptom score | Day 7 and day 14 of treatment initiation
  The secondary endpoints of the study include the statistical differences in the absolute values of changes in the Cough Severity Score (CSS) from baseline to Day 7 and Day 14 of treatment between the two groups of patients.
The change value of visual analog scale | Day 7 and day 14 of treatment initiation
  The secondary endpoints of the study include the statistical differences in the absolute values of changes in the Visual Analog Scale (VAS) score from baseline to Day 7 and Day 14 of treatment between the two groups of patients.
The change value of Athens Insomnia Scale | Day 7 and day 14 of treatment initiation
  The secondary endpoints of the study include the statistical differences in the absolute values of changes in the Airway Inflammation Score (AIS) from baseline to Day 7 and Day 14 of treatment between the two groups of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
All shared IPD will be de-identified to protect participant privacy, with direct identifiers (e.g., name, contact information, medical record numbers) removed or anonymized. Access to the data will be restricted to authorized researchers with a valid research proposal, ensuring the data is used only for purposes consistent with the original study's goals (e.g., secondary analyses of treatment efficacy or safety).